CLINICAL TRIAL: NCT03708822
Title: Open-Label, Multicenter, Phase Ⅱ Study of Docetaxel and Cisplatin Combined With Nimotuzumab As First-Line Treatment in Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma
Brief Title: Study of Docetaxel and Cisplatin Combined With Nimotuzumab As First-Line Treatment in Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2018-097-01
Record Dates: First submitted 2018-10-14; First posted 2018-10-17 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Docetaxel; Cisplatin; nimotuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Docetaxel and Cisplatin and Nimotuzumab (Experimental): All eligible patients received intravenous nimotuzumab plus docetaxel and cisplatin every 3 weeks for a maximum of 6 cycles, or until disease progression, death, intolerable toxicity.
  Interventions: Drug: Docetaxel and Cisplatin and Nimotuzumab

INTERVENTIONS:
Drug: Docetaxel and Cisplatin and Nimotuzumab — Intravenous nimotuzumab (200 mg on days 1, 8, and 15) ; Intravenous docetaxel (75 mg/m2 on day 1) ; Intravenous cisplatin (75 mg/m2 on day 1) ;

SUMMARY:
The purpose of this single arm,phase Ⅱ clinical trail is to determine the safety and efficacy of docetaxel and cisplatin combined with Nimotuzumab in the treatment of recurrent and metastatic nasopharyngeal carcinoma

ELIGIBILITY:
Inclusion Criteria:

* biopsy proved nasopharyngeal carcinoma;
* stage IVB according to the eighth edition American Joint Committee on Cancer/Union for International Cancer Control staging system, or recurrent disease beyond more than 6 months after curative chemotherapy and/or radiotherapy;
* 18-70 years;
* without other malignancy;
* had at least one measurable disease;
* had an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
* estimated life expectancy exceeding 3 months;
* adequate functions of the major organs.

Exclusion Criteria:

* allergic to docetaxel or cisplatin or nimotuzumab;
* pregnant or lactating female;
* patients received other clinical trails within 3 months;
* had serious infections, comorbidities or vital organs dysfunction.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
overall response rate | up to 18 weeks
  the proportion of patients achieved partial response (PR) and complete response (CR) according to RECIST v1.1

SECONDARY OUTCOMES:
disease control rate | up to 18 weeks
  the proportion of patients achieved CR, PR, or stable disease [SD]
duration of response | From date of documented response until the date of progressive disease [PD] or death, whichever came first, assessed up to 12 months
  time interval from the first day of documented response to progressive disease [PD] or death from any cause
progression-free survival | From date of the enrollment until the date of the documented PD or death, whichever came first, assessed up to 12 months
  time interval from the enrolled date to the documented PD or death from any cause or censored at the last follow-up
overall survival | From date of the enrollment until the date of the documented death, assessed up to 72 months
  time interval from the enrolled date to death from any cause or last follow-up
adverse events | up to 18 weeks
  treatment-related adverse events graded for severity according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University,, Guangzhou, China

REFERENCES:
- [Derived] Zou Q, Cao Y, Lai Y, Fang Y, Zhang Y, Liu P, Lu L, Wu H, Huang T, Su N, Li Z, Wang X, Tian X, Li L, Liu Y, Cai Q, Xia Y. Nimotuzumab combined with docetaxel and cisplatin as first-line treatment for patients with recurrent or metastatic nasopharyngeal carcinoma: a multicenter, phase 2 trial. BMC Med. 2025 May 6;23(1):264. doi: 10.1186/s12916-025-04103-0. PMID 40325445